CLINICAL TRIAL: NCT05133531
Title: A Randomized, Open-Label, C5 Inhibitor-Controlled Study to Evaluate the Efficacy and Safety of Pozelimab and Cemdisiran Combination Therapy in Patients With Paroxysmal Nocturnal Hemoglobinuria Who Are Complement Inhibitor Treatment-Naive or Have Not Recently Received Complement Inhibitor Therapy
Brief Title: A Study to Evaluate How Safe Pozelimab + Cemdisiran Combination Therapy is and How Well it Works in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Who Have Not Recently Received or Have Not Received Complement Inhibitor Treatment
Acronym: ACCESS-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-2021; 2020-004486-40 (EudraCT Number); 2023-509657-31-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab; eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Randomized 1:1
  Interventions: Drug: Ravulizumab; Drug: Pozelimab; Drug: Cemdisiran
- Cohort B (Experimental): Randomized 1:1
  Interventions: Drug: Pozelimab; Drug: Cemdisiran; Drug: Eculizumab

INTERVENTIONS:
Drug: Ravulizumab — Administered Intravenous (IV) per the protocol
  Other Names: ALXN1210; Ultomiris
  Arms: Cohort A
Drug: Pozelimab — Administered IV and subcutaneous (SC) per the protocol
  Other Names: REGN3918
Drug: Cemdisiran — Administered SC per the protocol
  Other Names: ALN-CC5
Drug: Eculizumab — Administered IV per the protocol
  Other Names: Soliris
  Arms: Cohort B

SUMMARY:
This study is researching a clinical treatment combination with two experimental drugs called pozelimab and cemdisiran. The study is focused on people with paroxysmal nocturnal hemoglobinuria (PNH). The aim of the study is to see how safe and effective the pozelimab + cemdisiran combination is for people with PNH and how the combination compares with 2 existing treatments: ravulizumab and eculizumab.

The pozelimab + cemdisiran combination may be referred to as "study drugs". Ravulizumab and eculizumab may also be called the "comparator drug".

The study is looking at several research questions, including:

* How effective is the pozelimab + cemdisiran combination compared to ravulizumab?
* How effective is pozelimab + cemdisiran combination compared to eculizumab?
* What side effects may happen from taking the study drugs?
* How much study drugs are in the blood at different times?
* Whether the body makes antibodies against the study drugs (which could make the study drugs less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of PNH confirmed by high-sensitivity flow cytometry testing with PNH granulocytes or monocytes as described in the protocol
2. Active disease, as defined by the presence of 1 or more PNH-related signs or symptoms as described in the protocol
3. LDH level ≥2 × ULN at the screening visit
4. Willing and able to comply with clinic/remote visits and study-related procedures, including completion of the full series of meningococcal vaccinations required per protocol

Key Exclusion Criteria:

1. Prior treatment with eculizumab within 3 months prior to screening, ravulizumab within 6 months prior to screening, or other complement inhibitors within 5 half-lives of the respective agent prior to screening
2. Receipt of an organ transplant, history of bone marrow transplantation or other hematologic transplant
3. Body weight <40 kilograms at screening visit
4. Planned use of any complement inhibitor therapy other than study drugs during the treatment period
5. Not meeting meningococcal vaccination requirements and, at a minimum documentation of quadrivalent meningococcal vaccination within 5 years prior to the screening visit and serotype B vaccine within 3 years prior to the screening visit as described in the protocol.
6. Any contraindication for receiving Neisseria meningitidis vaccinations (serotypes ACWY and B).
7. Unable to take antibiotics for meningococcal prophylaxis (if required by local ravulizumab [Cohort A] or eculizumab [Cohort B] prescribing information, where available, or national guidelines/local practice, or if necessary when administration of the first dose of the quadrivalent meningococcal vaccine [serotype ACWY] or the second dose of the serotype B meningococcal vaccine [when available] is less than 2 weeks prior to study treatment initiation) as described in the protocol
8. Any active, ongoing infection or a recent infection requiring ongoing systemic treatment with antibiotics, antivirals, or antifungals within 2 weeks of screening or during the screening period
9. Documented history of active, uncontrolled, ongoing systemic autoimmune diseases

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-01-28 (Estimated); Study Completion 2027-01-28 (Estimated)

PRIMARY OUTCOMES:
Percent change in lactate dehydrogenase (LDH) | From baseline to week 26
  Cohort A
Transfusion avoidance | From post-baseline day 1 through week 26
  Cohort B Not requiring a red blood cell (RBC) transfusion per the protocol
Adequate control of hemolysis | From week 8 through week 26, inclusive
  Cohort B LDH ≤1.5 × ULN at each visit

SECONDARY OUTCOMES:
Maintenance of adequate control of hemolysis | From week 8 through week 26, inclusive
  Cohort A and B LDH ≤1.5 × ULN
Breakthrough hemolysis | From post-baseline day 1 through week 26
  Cohort A and B LDH ≥2 × ULN per the protocol
Adequate control of hemolysis | From week 8 through week 26, inclusive
  Cohort A LDH ≤1.5 × ULN
Hemoglobin stabilization | From day 1 (post-baseline) through week 26
  Cohort A and B Patients who do not receive an RBC transfusion and have no decrease in hemoglobin level per the protocol
Normalization of LDH | Between week 8 through week 26, inclusive
  Cohort A and B LDH ≤1.0 × ULN per the protocol
Transfusion avoidance | Day 1 through week 26
  Cohort A Not requiring an RBC transfusion as per protocol algorithm based on post-baseline hemoglobin values.
Change in fatigue as measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale | From baseline to week 26
  Cohort A and B FACIT-Fatigue Scale is a 13-item, self-reported PRO measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related quality of life (QoL) in patients with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue.
Change in physical function (PF) scores on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) | From baseline to week 26
  Cohort A and B EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 7 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, sleep and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Change in global health status (GHS)/QoL scale score on the EORTC-QLC-C30 | From baseline to week 26
  Cohort A and B EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 7 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, sleep and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Percent change in LDH | From baseline to week 26
  Cohort B
Rate of RBC transfused | Post-baseline Day 1 through week 26
  Cohort A and B Per protocol algorithm
Number of units of RBC transfused | Post-baseline Day 1 through week 26
  Cohort A and B Per protocol algorithm
Time to first LDH ≤1.5 × ULN | Up to Week 26
  Cohort A and B
Time to first LDH ≤1.0 × ULN | Up to Week 26
  Cohort A and B
Percentage of days with LDH ≤1.5 × ULN | Between week 8 and week 26, inclusive
  Cohort A and B
Change in hemoglobin levels | From baseline to week 26
  Cohort A and B
Incidence and severity of treatment emergent serious adverse events (SAEs) | Up to 26 weeks
  Cohort A and B
Incidence and severity of treatment-emergent adverse events (TEAEs) of special interest | Up to 26 weeks
  Cohort A and B
Incidence and severity of TEAEs leading to treatment discontinuation | Up to 26 weeks
  Cohort A and B
Change in total CH50 | From baseline to week 26
  Cohort A and B
Percent change in total CH50 | From baseline to week 26
  Cohort A and B
Concentration of total C5 in plasma | Up to 60 weeks
  Cohort A and B
Concentrations of total pozelimab in serum | Up to 60 weeks
  Cohort A and B
Concentrations of cemdisiran in plasma | Up to 60 weeks
  Cohort A and B
Concentrations of total ravulizumab in serum | Up to 34 weeks
  Cohort A
Concentrations of total eculizumab in serum | Up to 30 weeks
  Cohort B
Incidence of treatment emergent anti-drug antibodies (ADAs) to pozelimab | Up to 60 weeks
  Cohort A and B
Incidence of treatment emergent ADAs to cemdisiran | Up to 60 weeks
  Cohort A and B

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (69):
- The Oncology Institute of Hope & Innovation, Whittier, California, United States
- Brazil (3):
  - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André, São Paulo
  - A Beneficencia Portuguesa de Sao Paulo, BP Mirante, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo
- Toronto General Hospital, Toronto, Ontario, Canada
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China
- Hospital Pablo Tobon Uribe, Medellín, Antioquia, Colombia
- George Papanikolaou Hospital, Thessaloniki, Greece
- Semmelweis University, Budapest, Hungary
- India (8):
  - Malabar Cancer Center, Kerala, Kannur, Kerala
  - Amrita Institute of Medical Sciences (AIMS) and Research Centre Aims, Kochi, Kerala
  - K J Somaiya Super Specialty Hospital & Research Centre, Mumbai, Maharashtra
  - Rajiv Gandhi Cancer Institute & Research Center (RGCIRC) - Rohini Campus, New Delhi, National Capital Territory of Delhi
  - Postgraduate Institute of Medical Education & Research (PGIMER), Chandigarh, Punjab
  - King George Hospital, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Bhagwan Mahaveer Cancer Hospital and Research Centre (BMCHRC), Jaipur
- Italy (3):
  - Aou Careggi, Florence, Firenze
  - Fondazione Policlinico Universitrio a. Gemelli - IRCCS, Rome, Roma
  - Hematology Citta della Salute e della Scienza di Torino, Turin
- Japan (5):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Matsushita Memorial Hospital, Moriguchi, Osaka
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
- Jordan University Hospital (JUH), Amman, Jordan
- Malaysia (3):
  - Hospital Tg Ampuan Afzan, Kuantan, Pahang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
- Servicio de Hematologia del Hospital Universitario de la Uanl, Monterrey, Nuevo León, Mexico
- Clinica San Felipe, Lima, Peru
- St Lukes Medical Center, Quezon, Central Luzon, Philippines
- Poland (3):
  - University Clinical Center Medical University of Gdansk, Gdansk, Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr2 Bydgoszcz, Bydgoszcz
  - Institute of Hematology and Transfusion Medicine, Warsaw
- Romania (3):
  - Ion Chiricuta Oncology Institute, Cluj-Napoca, Cluj
  - Municipal Hospital Filantropia, Craiova, Dolj
  - Targu Mures Clinical County Emergency Hospital, Târgu Mureş, Mureș County
- National University Hospital, Singapore, Singapore
- South Korea (9):
  - St. Vincent Hospital, Suwon, Gyeonggi-do
  - Ajou University Medical Center, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Namdong-Gu
  - Pusan National University Hospital, Busan
  - Korea University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital - The Catholic University of Korea, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (4):
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General JM Morales Meseguer, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Taiwan (9):
  - China Medical University Hospital, Taichung, Central Taiwan
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District, Hunan Province
  - Changhua Christian Hospital, Changhua
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital (VGHTC), Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (5):
  - Clinical Research Center, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Chaing Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul
  - Ege University, Izmir
- St James Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry),
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: Study Informational Website — https://access1study.com/